CLINICAL TRIAL: NCT06155058
Title: Comparison Of Robotic And Conventional Mirror Therapy On Hand Motoric Recovery And Functional Outcomes For Rehabilitation Of Post-Stroke Patients
Brief Title: Robotic Versus Conventional Therapy For Post-Stroke Hand Motoric Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Bumi Herman, Assistant Lecturer, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2411232122
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Stroke; Physical Disability; Upper Extremity Paresis
Keywords: Robotic Therapy; Mirror Therapy; Post-Stroke; Upper Extremities; Motoric Function; Functional Outcome
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Intervention Model Description: The intervention group will be the robotic and the active comparator will be the conventional mirror therapy exercise group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Mirror Therapy (Experimental): Serial training with the help of exoskeletal robot therapy
  Interventions: Procedure: SYREBO
- Conventional Mirror Therapy (Active Comparator): Serial training with the help of physical therapist
  Interventions: Procedure: Conventional Mirror Method

INTERVENTIONS:
Procedure: SYREBO — Serial ADL training of upper extremities with robotic aid
  Arms: Robotic Mirror Therapy
Procedure: Conventional Mirror Method — Serial ADL training of upper extremities assisted by physical therapist
  Arms: Conventional Mirror Therapy

SUMMARY:
This clinical trial aims to compare the effectiveness of Robotic versus conventional mirror therapy among post-stroke patients. The main questions it aims to answer are:

* Effectiveness of both interventions in hand motoric recovery across time
* Effectiveness of both interventions in functional outcomes across time
* Clinical outcome difference between both interventions Participants will be allocated into either a robotic group as the main intervention or a mirror therapy group as the active comparator. A serial follow-up will be conducted to assess the selected clinical outcome and differences in outcome

DETAILED DESCRIPTION:
1. Research design This research is an experimental study with a randomized controlled trial research design.
2. Study Setting The research will be carried out among post-stroke patients at two teaching hospitals and one physical rehabilitation centre in Makassar
3. Procedure

   1. Robotic Procedure an exoskeletal robot (Syrebo) will help and stimulate the movement of the paralyzed extremity. One set of training covering Activity Daily Living (ADL) set will be conducted. A mirror will reflect the movement of the healthy extremities
   2. Conventional Method the difference from the robotic procedure was, the movement and stimulation will be provided by the physical therapist.
4. Time frame the procedure will be conducted in parallel three times per week for a total of six weeks
5. Outcomes

   1. motoric ability of upper extremity using Fugl-Meyer Assessment for Upper Extremities (FMA-UE)
   2. Dexterity, coordination and response of finger using the Nine Hole Peg Test (NHPT)
6. Covariates and potential confounders

   1. type of stroke determined by radiology imaging
   2. phase of stroke (acute, sub-acute or chronic)
   3. cognitive ability measured using mini-mental state examination (MMSE)
   4. Spasticity measured by the Modified Ashworth Scale (MAS)
7. Procedure The data collected is primary data obtained in accordance with the inclusion criteria.

   Samples who are willing to become research subjects will undergo interviews, physical examinations, FMA-UE-Hand Motor Domain and NHPT examinations. The interview questionnaire in this study will contain a list of patient identities including name, age, marital status, address, educational history, employment history, history of stroke, cognitive examination (MMSE), and self-reported visual ability.

   The FMA-UE-Hand Motor Domain scoring system is used to evaluate upper extremity motor function in patients with neurological disorders, such as stroke. The scoring system ranges from 0-14, with higher scores indicating better motor function. The FMA-UE-Hand Motor domain assessment system is broken down into several subscales, namely Mass Flexion and Extension movements, followed by functional movements of grasping (Grasp), including Hook Grasp, Thumb Adduction, Pincer Grasp, Cylinder Grasp, and Spherical Grasp. The assessment will get a score of 0 = None or no movement, 1 = Partial or limited movement, and 2 = Full or perfect movement.

   The NHPT assessment consists of a square board with 9 pegs. At one end of the board, there is a hole for the peg, and at the other end, there is a shallow round plate for holding the peg. NHPT is performed by having the patient take pegs from a container, one at a time, and place them into the holes in a board, as quickly as possible. The patient must then remove the pegs from the holes, one at a time, and reinsert them into the housing. To practice and register initial scores, the test must be started with the unaffected upper limb. The board should be placed in the centre of the patient's body with the housing holding the pegs oriented toward the hand being tested. Only the hand being evaluated should perform the test. The non-evaluated hand is allowed to grip the edge of the board to provide stability. Patients are scored based on the time required to complete the test activity, recorded in seconds. The stopwatch must start from the moment the participant touches the first peg until the last peg touches the container. This assessment requires a board, of wood or plastic, with 9 holes (10 mm diameter, 15 mm depth), spaced 32 mm or 50 mm apart and a stopwatch.
8. Sample Size Based on previous research, the value of the standard deviation of the selected outcome = 11.5 and the value of x1-x2 = 9.1 (Lin, 2020). The Zα value = 1.96 with a confidence interval of 95% and the Zβ value = 0.84 with a power of 80%, two arms and a dropout rate of 30% at least 40 participants should be recruited. A consecutive sampling will be applied and allocated randomly using the simple randomization technique.
9. Proposed Statistical Analysis Data on the effect of robotic mirror therapy compared to conventional mirror therapy will be assessed using the independent t-test. Data from the FMA-UE and NHPT assessments before and after the intervention will be analyzed using the paired t-test. Next, the relationship between the FMA-UE and NHPT values will be assessed using the Pearson correlation test (normally distributed data) or the Spearman test (data not normally distributed) to determine how big the correlation is between these variables.

ELIGIBILITY:
Inclusion criteria:

1. Patients aged 20 - 85 years.
2. Non-haemorrhagic stroke/infarction with onset more than 3 months from the onset of the attack.
3. Patients with unilateral upper limb hemiparesis.
4. Modified Ashworth Scale (MAS) on fingers and hands <3
5. The patient has not undergone mirror therapy treatment before.
6. Patients who are able to understand informed consent to participate in research.
7. The patient had a Radiology imaging of the head at the time of stroke onset.

Exclusion criteria:

1. Patients with severe spasticity or contractures of the upper extremities.
2. Patients with infarction/bleeding with extensive lesions covering 2 hemispheres.
3. The patient has severe cognitive impairment that will interfere with the research objectives (MMSE score >24).
4. Patients post Digital Subtraction Angiography (DSA) procedures in the last 2 months.
5. Patients with a history of seizures or epilepsy.
6. Patients with visual field deficits or severe visual impairment.
7. Patients who are unable to sit upright without assistance.
8. Other uncontrolled medical conditions (musculoskeletal, neuromuscular, cardiorespiratory) that may interfere with the ability to exercise.

Dropout criteria:

Patients were excluded from the study if:

1. Participant dies.
2. Participants take part in the exercise <3 times for 2 consecutive weeks.
3. The participant refuses to continue the training session.
4. Participants experience hemodynamic disorders during the training program phase.
5. Participants experience neurological disorders during the training program phase.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
FMA-UE Score | changes of FMA-UE score from pre-intervention to six weeks after intervention
  a motoric assessment with each score range from 0-2 with a total score range from 0-66. Higher score indicates better and free movement
NHPT value | changes of NHPT values from pre-intervention to six weeks after intervention
  an assessment for finger dexterity and coordination where the time of the subject to accomplish task will be recorded. Average healthy adult male completed the NHPT in 19.0 seconds (SD 3.2) with the right hand, and in 20.6 seconds (SD 3.9) with the left hand. For healthy adult women, the NHPT was completed in 17.9 seconds (SD 2.8) and 19.6 seconds (SD 3.4) with the right and left hands, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kurniawan, MD, Principal Investigator — Hasanuddin University; Nuralam Sam, MD. Ph.D, Principal Investigator — Hasanuddin University; Husnul Mubarak, MD, Principal Investigator — Hasanuddin University; Yose Waluyo, MD. PhD, Principal Investigator — Hasanuddin University; Andi A Zainuddin, MD.Phd, Principal Investigator — Hasanuddin University; Andi A Mochtar, Dr. Eng, Principal Investigator — Hasanuddin University
Locations (3):
- Indonesia (3):
  - Cerebellum Clinic, Makassar, South Sulawesi
  - Hasanuddin University, Faculty of Medicine, Makassar, South Sulawesi
  - Wahidin Sudirohusodo General Hospital, Makassar, South Sulawesi

IPD SHARING:
Plan to Share IPD: No
To protect the confidentiality, should the data need to share, any de-identified data will be shared for peer-review

REFERENCES:
- [Background] Beom J, Koh S, Nam HS, Kim W, Kim Y, Seo HG, Oh BM, Chung SG, Kim S. Robotic Mirror Therapy System for Functional Recovery of Hemiplegic Arms. J Vis Exp. 2016 Aug 15;(114):54521. doi: 10.3791/54521. PMID 27583794
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Chowdhury, Z., 2018. Effectiveness of Mirror Therapy on hand function improvement among patients with chronic stroke. IOSR Journal of Nursing and Health Science (IOSR-JNHS) e-ISSN: 2320-1959.p- ISSN: 2320-1940 Volume 4, Issue 6 Ver. V (Nov. - Dec. 2015), PP 01-04
- [Background] Hijikata N, Kawakami M, Ishii R, Tsuzuki K, Nakamura T, Okuyama K, Liu M. Item Difficulty of Fugl-Meyer Assessment for Upper Extremity in Persons With Chronic Stroke With Moderate-to-Severe Upper Limb Impairment. Front Neurol. 2020 Nov 16;11:577855. doi: 10.3389/fneur.2020.577855. eCollection 2020. PMID 33304304
- [Background] Lee MM, Cho HY, Song CH. The mirror therapy program enhances upper-limb motor recovery and motor function in acute stroke patients. Am J Phys Med Rehabil. 2012 Aug;91(8):689-96, quiz 697-700. doi: 10.1097/PHM.0b013e31824fa86d. PMID 22469877
- [Background] Nogueira NGHM, Parma JO, Leao SESA, Sales IS, Macedo LC, Galvao ACDR, de Oliveira DC, Murca TM, Fernandes LA, Junqueira C, Lage GM, Ferreira BP. Mirror therapy in upper limb motor recovery and activities of daily living, and its neural correlates in stroke individuals: A systematic review and meta-analysis. Brain Res Bull. 2021 Dec;177:217-238. doi: 10.1016/j.brainresbull.2021.10.003. Epub 2021 Oct 7. PMID 34626693
- [Background] Rothgangel AS, Braun SM, Beurskens AJ, Seitz RJ, Wade DT. The clinical aspects of mirror therapy in rehabilitation: a systematic review of the literature. Int J Rehabil Res. 2011 Mar;34(1):1-13. doi: 10.1097/MRR.0b013e3283441e98. PMID 21326041
- [Background] Schrader M, Sterr A, Kettlitz R, Wohlmeiner A, Buschfort R, Dohle C, Bamborschke S. The effect of mirror therapy can be improved by simultaneous robotic assistance. Restor Neurol Neurosci. 2022;40(3):185-194. doi: 10.3233/RNN-221263. PMID 35848045